CLINICAL TRIAL: NCT03092895
Title: A Phase 2 Study of SHR-1210 (PD-1 Antibody) in Combination With Apatinib or Chemotherapy (FOLFOX4 or GEMOX) in Subjects With Advanced Primary Liver Cancer（PLC）or Biliary Tract Carcinoma (BTC)
Brief Title: A Study of SHR-1210 in Combination With Apatinib or Chemotherapy in Subjects With Advanced PLC or BTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-APTN-II-203-PLC
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2022-04

CONDITIONS: Advanced Primary Liver Cancer; Advanced Biliary Tract Carcinoma
MeSH Terms: interventions — camrelizumab; apatinib; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210+Apatinib(Arm A） (Experimental)
  Interventions: Biological: SHR-1210; Drug: Apatinib
- SHR-1210+FOLFOX4 or GEMOX regimen(Arm B） (Experimental)
  Interventions: Biological: SHR-1210; Drug: FOLFOX4; Drug: GEMOX

INTERVENTIONS:
Biological: SHR-1210 — Subjects receive SHR-1210 intravenous at the dose 3mg/kg on Day 1 every 2 weeks
Drug: Apatinib — Subjects receive Apatinib orally every day with a dose escalation
  Arms: SHR-1210+Apatinib(Arm A）
Drug: FOLFOX4 — Subjects receive FOLFOX4 treatment every 2 weeks
  Arms: SHR-1210+FOLFOX4 or GEMOX regimen(Arm B）
Drug: GEMOX — Subjects receive GEMOX treatment every 2 weeks
  Arms: SHR-1210+FOLFOX4 or GEMOX regimen(Arm B）

SUMMARY:
This an open-label，Non-Randominzed Phase 2 study to evaluate the Safety and Tolerability of SHR-1210 in combination with Apatinib or chemotherapy (FOLFOX4 or GEMOX regimen) in subjects with Advanced PLC.or BTC Participants with advanced PLC who failed or intolerable to prior systemic therapy will be treated with SHR-1210 plus Apatinib; Participants with advanced PLC or BTC who have never received prior systemic therapy will be treated with SHR-1210 plus FOLFOX4 or GEMOX regimen.

ELIGIBILITY:
1. Histologically confirmed advanced PLC or advanced BTC (including bile duct carcinoma and gallbladder carcinoma) ; not suitable to surgery or local regional treatment; with at least one measurable lesion per RECIST 1.1.
2. Arm A:Failed or intolerable to at least one prior systemic treatment for advanced PLC. Arm B:No previous systemic treatment for advanced PLC or BTC
3. ECOG Performance Status of 0 or1.
4. Child-Pugh Class A or B with 7 points .
5. Life Expectancy of at least 12 weeks.
6. Has controlled infection by Hepatitis B Virus (HBV DNA<500 IU/ml) or Hepatitis C Virus.
7. Adequate organ function.
8. Male or female participants of childbearing potential must be willing to use an adequate method of contraception starting with the first dose of study drug through 60 days for female subjects and 120 days for male subjects after the last dose of study drug.
9. Patient has given written informed consent.

Exclusion Criteria:

1. Known fibrolamellar HCC; Prior malignancy active with the previous 5 years except for locally curable cancers that have been apparently cured.
2. Known or occurrence of central nervous system (CNS) metastases.
3. Ascites with clinical symptoms.
4. Known or evidence of GI hemorrhage within the past 6 months.
5. Known or occurrence of hemorrhage/ thrombus.
6. Known or evidence of abdomen fistula, gastrointestinal perforation, or abdominal abscess within the past 2 months.
7. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias.
8. Grade III~IV cardiac insufficiency, according to NYHA criteria or echocardiography check: LVEF<50%.
9. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents (systolic blood pressure > 140mmHg, diastolic blood pressure > 90 mmHg).
10. Factors to affect oral administration (such as patients unable to swallow oral medications, chronic diarrhea and ileus etc. situations evidently affect drug oral medication and absorption).
11. History of hepatic encephalopathy.
12. Known history of human immunodeficiency virus (HIV) infection.
13. Active infection or an unexplained fever > 38.5°C during screening visits.
14. Has received a live vaccine within 30 days.
15. Prior or planning to organ transplantation including liver transplantation.
16. Interstitial lung disease that is symptomatic or may interfere with the detection and management of suspected drug-related pulmonary toxicity.
17. Proteinuria≥ 2+ or 24 hours total urine protein > 1.0 g.
18. Active known, or suspected autoimmune disease.
19. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily. prednisone equivalent, are permitted in the absence of active autoimmune disease
20. Any loco-regional therapy to liver (included but not limited: resection, radiotherapy, TAE, TACE, TAI, RFA or PEI) within 4 weeks prior to study.
21. Prior therapy with anti-PD-1 or other anti-PD-1/anti-PD-L1 immunotherapy.
22. Known history of hypersensitivity to monoclonal antibodies or any components of the study drugs.
23. Treatment with anti-coagulation therapy(Warfarin or heparin) or anti-platelet therapy(aspirin at dose≥300mg/day, clopidogrel at dose≥75mg/day).
24. Pregnant or breast-feeding women.
25. According to the investigator, other conditions that may lead to stop the research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - The Second Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Hunan Cancer Hospital, Hunan, Changsha
  - Cancer Hospital of Henan province, Zhengzhou, Henan
  - 81 Hospital Nanjing, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Jiangxi, Nanchang
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Qin S, Gu S, Ren Z, Chen Z, Xiong J, Liu Y, Meng Z, Zhang X, Wang L, Zhang X, Zou J. Camrelizumab plus oxaliplatin-based chemotherapy as first-line therapy for advanced biliary tract cancer: A multicenter, phase 2 trial. Int J Cancer. 2021 Dec 1;149(11):1944-1954. doi: 10.1002/ijc.33751. Epub 2021 Sep 8. PMID 34309846
- [Derived] Mei K, Qin S, Chen Z, Liu Y, Wang L, Zou J. Camrelizumab in combination with apatinib in second-line or above therapy for advanced primary liver cancer: cohort A report in a multicenter phase Ib/II trial. J Immunother Cancer. 2021 Mar;9(3):e002191. doi: 10.1136/jitc-2020-002191. PMID 33741732

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A：SHR-1210+Apatinib: SHR-1210: 3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days.
  Apatinib mesylate: Orally administered, once daily, with four dose groups: 125 mg, 250 mg, 375 mg, and 500 mg, for dose exploration from low dose to high dose.
- Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W): SHR-1210 + FOLFOX4 Q2W： SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days； FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
- Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W); Arm B：Others: SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W:D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
Period: Overall Study
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others
Started | 28 | 34 | 92 | 3
Completed | 28 | 34 | 92 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W): SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
- Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W): SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W：D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
- Arm B：Others: SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W： D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others | Total
Number analyzed (Participants) | 28 | 34 | 92 | 3 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (9.77) | 52.2 (8.75) | 53.9 (9.71) | 53.0 (13.00) | 52.9 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 37 | 2 | 49
  Male | 21 | 31 | 55 | 1 | 108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability
Description: The incidence of adverse events (AEs) and Serious adverse events (SAEs) assessed by NCI-CTCAE v4.03
Time Frame: Up to approximately 4 years
Population: The primary safety endpoint was analyzed in SS. The SS included all participants who were treated .
Measure: Number; unit: participants
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
participants
  Number of Subjects with AEs | 28 | 34 | 92 | 3
  Number of Subjects with SAEs | 14 | 20 | 58 | 2

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) assessed by investigator: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm B：Hepatocellular Carcinoma(SHR-1210+ FOLFOX4 Q2W): SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
- Arm B：Others: SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W：D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210+ FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
percentage of participants | 10.7 [2.3 to 28.2] | 29.4 [15.1 to 47.5] | 16.3 [9.4 to 25.5] | 33.3 [0.8 to 90.6]

3. Secondary Outcome: Duration of Response (DoR)
Description: The time from the date of the first recorded objective tumor response (assessed as per RECIST V1.1) to the date of the first recorded objective tumor progression (assessed as per RECIST V1.1) or the date of death due to any cause, whichever occurs first, in subjects with a BOR of CR or PR.
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Median (Full Range); unit: months
Groups:
- Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W); Arm B：Others: SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days；
  FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W： D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
months | 11.30 [11.3 to 11.3] | 7.10 [3.3 to 29.7] | 7.10 [3.6 to 20.2] | 7.20 [7.2 to 7.2]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of subjects with a BOR of CR, PR, and SD as per RECIST V1.1. BOR of CR or PR must be confirmed at least 4 weeks (28 days) after the initial assessment.
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210+ GEMOX Q2W); Arm B：Others: SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days； FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W： D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210+ GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
percentage of participants | 64.3 [44.1 to 81.4] | 79.4 [62.1 to 91.3] | 75.0 [64.9 to 83.4] | 33.3 [0.8 to 90.6]

5. Secondary Outcome: Time to Progression (TTP)
Description: The time from the date of the first dose to the date of radiographic PD (assessed by the investigator as per RECIST V1.1).PD is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or significant progression of non-target lesions leading to discontinuation of therapy, or the appearance of new lesions.
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210+ FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210+ GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
months | 3.7 [2.0 to 5.7] | 5.7 [3.8 to 9.2] | 5.5 [3.7 to 7.3] | 2.0 [1.8 to NA] — not reached (due to insufficient number of subjects with events).

6. Secondary Outcome: Overall Survival
Description: The time from the date of the first dose to death due to any cause. Overal Survial will be calculated based on Kaplan-Meier estimates
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm B：Cholangiocarcinoma（SHR-1210+ FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W): SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days； FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W：D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210+ FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
months | 13.3 [8.9 to 18.6] | 11.7 [8.2 to 19.0] | 10.7 [7.7 to 15.4] | 17.6 [4.8 to NA] — not reached (due to insufficient number of subjects with events)

7. Secondary Outcome: Time to Response (TTR)
Description: The time from the date of the first dose to the date of the first recorded tumor response (assessed as per RECIST V1.1) in subjects with a BOR of CR or PR.
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Median (Full Range); unit: months
Groups:
- Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210+ GEMOX Q2W); Arm B：Others: SHR-1210：3 mg/kg, intravenously infused within 30 min, not less than 20 min and not more than 60 min (including flushing time), once every 2 weeks. The interval between two doses must not be less than 12 days； FOLFOX4 regimen：D1: Oxaliplatin (OXA) 85 mg/m2 (2-h infusion) + calcium levofolinate (LV) 200 mg/m2 (2-h infusion), followed by 5-fluorouracil (5-Fu) 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion)，D2: LV 200 mg/m2 (2-h infusion), followed by 5-Fu 400 mg/m2 (bolus injection), and 5-Fu 600 mg/m2 (22-h infusion) Once every 2 weeks.
  GEMOX Q2W：D1: Gemcitabine (800 mg/m2, 80-min infusion) ，D2: Oxaliplatin (85 mg/m2, 2-h infusion) Once every 2 weeks.
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210+ FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210+ GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
months | 3.65 [1.8 to 3.7] | 1.99 [1.5 to 5.6] | 1.84 [1.7 to 5.7] | 1.87 [1.87 to 1.87]

8. Secondary Outcome: Progression-free Survival (PFS)
Description: The time from the date of the first dose to the date of the first recorded tumor progression (assessed as per RECIST V1.1) or the date of death due to any cause, whichever occurs first.
Time Frame: Up to approximately 4 years
Population: The secondary efficacy endpoint was analyzed in FAS. The FAS included all participants who were treated.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210+ GEMOX Q2W) | Arm B：Others
Number analyzed (Participants) | 28 | 34 | 92 | 3
months | 3.7 [2.0 to 5.7] | 5.7 [3.8 to 9.2] | 5.3 [3.7 to 5.7] | 2.0 [1.8 to NA] — not reached (due to insufficient number of subjects with events).

ADVERSE EVENTS:
Time Frame: Up to approximately 4 years
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Arm A：SHR-1210+Apatinib | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) | Arm B：Others
All-Cause Mortality (participants affected / at risk) | 11/28 | 11/34 | 35/92 | 1/3
Serious Adverse Events (participants affected / at risk) | 14/28 | 20/34 | 58/92 | 2/3
Other Adverse Events (participants affected / at risk) | 28/28 | 34/34 | 92/92 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A：SHR-1210+Apatinib (N=28) | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) (N=34) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) (N=92) | Arm B：Others (N=3)
Hepatic failure (Hepatobiliary disorders) | 4 | 3 | 7 | 0
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 3 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 3 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 3 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 5 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 4 | 7 | 1
Disease progression (General disorders) | 0 | 2 | 10 | 0
Pyrexia (General disorders) | 0 | 1 | 7 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 4 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 7 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 2 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4 | 2 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 3 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Reactive capillary endothelial proliferation (Immune system disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 2 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Eating disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A：SHR-1210+Apatinib (N=28) | Arm B：Hepatocellular Carcinoma(SHR-1210 + FOLFOX4 Q2W) (N=34) | Arm B：Cholangiocarcinoma（SHR-1210 + FOLFOX4 Q2W or SHR-1210 + GEMOX Q2W) (N=92) | Arm B：Others (N=3)
Anaemia (Blood and lymphatic system disorders) | 6 | 13 | 45 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 6 | 0
Hypothyroidism (Endocrine disorders) | 8 | 5 | 14 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 2 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 8 | 24 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 10 | 25 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 15 | 1
Vomiting (Gastrointestinal disorders) | 5 | 7 | 40 | 1
Constipation (Gastrointestinal disorders) | 4 | 10 | 26 | 1
Nausea (Gastrointestinal disorders) | 4 | 9 | 25 | 3
Stomatitis (Gastrointestinal disorders) | 4 | 1 | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 13 | 1
Ascites (Gastrointestinal disorders) | 3 | 7 | 11 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 7 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 3 | 1 | 6 | 0
Abdominal pain lower (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 4 | 0
Noninfective gingivitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 10 | 9 | 33 | 1
Pyrexia (General disorders) | 9 | 10 | 56 | 2
Chest discomfort (General disorders) | 3 | 1 | 4 | 0
Face oedema (General disorders) | 2 | 1 | 8 | 0
Oedema peripheral (General disorders) | 1 | 2 | 10 | 1
Reactive capillary endothelial proliferation (Immune system disorders) | 6 | 26 | 57 | 3
Aspartate aminotransferase increased (Investigations) | 23 | 22 | 53 | 2
Platelet count decreased (Investigations) | 22 | 30 | 49 | 2
Bilirubin conjugated increased (Investigations) | 20 | 15 | 18 | 2
Blood bilirubin increased (Investigations) | 19 | 16 | 28 | 2
White blood cell count decreased (Investigations) | 18 | 30 | 49 | 3
Neutrophil count decreased (Investigations) | 17 | 29 | 44 | 3
Alanine aminotransferase increased (Investigations) | 15 | 14 | 43 | 0
Gamma-glutamyltransferase increased (Investigations) | 10 | 10 | 37 | 1
Weight decreased (Investigations) | 10 | 6 | 21 | 0
Blood lactate dehydrogenase increased (Investigations) | 7 | 8 | 15 | 2
Blood alkaline phosphatase increased (Investigations) | 6 | 13 | 35 | 0
Haemoglobin decreased (Investigations) | 5 | 2 | 7 | 2
Weight increased (Investigations) | 5 | 7 | 8 | 0
Blood albumin decreased (Investigations) | 4 | 5 | 6 | 1
Blood bilirubin unconjugated increased (Investigations) | 4 | 2 | 3 | 0
Blood thyroid stimulating hormone increased (Investigations) | 4 | 0 | 0 | 0
Amylase increased (Investigations) | 3 | 7 | 10 | 1
Hepatitis B DNA increased (Investigations) | 3 | 0 | 0 | 0
Lipase increased (Investigations) | 3 | 9 | 19 | 1
Albumin globulin ratio decreased (Investigations) | 2 | 2 | 3 | 0
Blood creatinine increased (Investigations) | 2 | 1 | 10 | 1
Blood glucose increased (Investigations) | 2 | 2 | 4 | 0
Blood pressure increased (Investigations) | 2 | 1 | 5 | 0
Urobilinogen urine increased (Investigations) | 2 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 1 | 2 | 4 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 8 | 0
Red blood cell count decreased (Investigations) | 1 | 3 | 5 | 1
White blood cell count increased (Investigations) | 1 | 0 | 10 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 15 | 33 | 1
Decreased appetite (Metabolism and nutrition disorders) | 9 | 15 | 41 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 7 | 27 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 7 | 12 | 14 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 1 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3 | 19 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1 | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 10 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 8 | 1
Headache (Nervous system disorders) | 5 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 3 | 6 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 7 | 6 | 0
Insomnia (Psychiatric disorders) | 3 | 1 | 7 | 1
Proteinuria (Renal and urinary disorders) | 14 | 7 | 13 | 0
Haematuria (Renal and urinary disorders) | 5 | 4 | 6 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 11 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 10 | 1
Hypertension (Vascular disorders) | 22 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 3 | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 2 | 3 | 0
Chills (General disorders) | 0 | 1 | 11 | 0
Temperature intolerance (General disorders) | 0 | 0 | 5 | 0
Hypersensitivity (Immune system disorders) | 0 | 6 | 14 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 7 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 7 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1
Total bile acids increased (Investigations) | 0 | 1 | 7 | 0
Myoglobin blood increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil percentage decreased (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 6 | 0
Neurotoxicity (Nervous system disorders) | 0 | 3 | 1 | 1
Dysphoria (Psychiatric disorders) | 0 | 0 | 1 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 0
Phlebitis (Vascular disorders) | 0 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-05-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT03092895/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03092895/SAP_001.pdf